CLINICAL TRIAL: NCT00504985
Title: Fatigue and Its Symptom Cluster Related to Inflammatory Cytokine Profiles in Cancer Patients Seeking Emergency Care
Brief Title: Fatigue in Emergency Center Patients
Status: Terminated | Type: Observational
Why Stopped: Low Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2005-0266
Record Dates: First submitted 2007-07-18; First posted 2007-07-20 (Estimated); Results first posted 2010-05-04 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Advanced Cancer; Hematologic Malignancy; Fatigue
Keywords: Advanced Cancer; Hematologic Malignancy; Fatigue; Emergency Center; Survey
MeSH Terms: conditions — Hematologic Neoplasms; Fatigue | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — About 1 tablespoon of blood drawn for cytokine testing.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fatigue in Emergency Center Patients
  Interventions: Behavioral: Surveys

INTERVENTIONS:
Behavioral: Surveys — 2 surveys, taking about 10-15 minutes each, during Emergency Center visit
  Other Names: Questionniare

SUMMARY:
1. To describe fatigue severity and its related symptom clusters in cancer patients who are seeking emergency care for fever, pain, shortness of breath, or cancer therapy-related gastrointestinal toxicities.
2. To describe inflammatory cytokine profiles in cancer patients who are seeking emergency care for fever, pain, shortness of breath, or cancer therapy-related gastrointestinal toxicities.
3. To determine the type of cytokines that are associated with fatigue severity in cancer patients, with or without cancer treatment, in the early phase of infection, as well as in patients with pain, shortness of breath, or cancer therapy-related gastrointestinal toxicities.

DETAILED DESCRIPTION:
One of the ways to learn about the symptoms of cancer and the effect of cancer treatment is by rating how severe symptoms are and how they interfere with daily activity. Researchers can also compare these ratings to the levels of certain proteins called cytokines that are found in the blood while the patient is experiencing symptoms.

If you agree to take part in this study, you will be asked to complete 2 surveys during your Emergency Center visit. One survey will measure physical and mental symptoms (such as sadness or distress). The other survey will ask you for personal "demographic" information (such as your age and marital status). Completing the questionnaires will take about 10-15 minutes. During the Emergency Center visit, about 1 tablespoon of blood will be drawn for cytokine testing.

Research staff will also collect other information from your medical record, clinical information, and lab results. This information may include cancer diagnosis, cancer treatment, performance status (your ability to perform daily activities), disease status, and any medications you are taking at that time.

This is an investigational study. About 520 patients will participate in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be admitted to the Emergency Center with a diagnosis of cancer confirmed by pathology (either hematologic malignancies or solid tumors).
2. Patients with either hematologic malignancies or solid tumors must either be currently undergoing active cancer treatment (received chemotherapy, radiotherapy, chemoradiotherapy, blood or bone morrow transplant, surgery, immunotherapy anytime during the past month) or not receiving any cancer treatments in past month.
3. Patient's chief complaint upon admission to the EC must be one or more of the following four conditions: a. fever (38.3°C or higher) in past 24 hours b. pain c.any chemotherapy-related GI toxicities (such as nausea, vomiting, diarrhea, or constipation) d.shortness of breath
4. Patients must be able to read and write English
5. Patients must agree to participate and must sign the Informed Consent
6. Patients must be 18 years or older (minimal numbers of children are evaluated in the EC)
7. Patients must be able to complete the survey tool independently (without input or influence from their caregivers).
8. Patients whose performance status allows them to complete the survey (i.e., patients who do not have altered mental/cognitive status, and patients without emergent illness and hemodynamic instability---for example, status epilepticus, sepsis, cardiac arrest, and any life-threatening condition).

Exclusion Criteria:

1) Patients who were already enrolled on this protocol in a previous visit to this EC will not be enrolled again, regardless of their reasons for the current EC visit (same or different reason).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients admitted to the UT MD Anderson Cancer Center Emergency Center who are seeking emergency care for fever, pain, shortness of breath, or cancer therapy-related gastrointestinal toxicities.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2005-08; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xin Shelley Wang, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 07/19/06 through 10/18/06. All participants recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Study terminated early due to low accrual.
Period: Overall Study
Arm/Group | Fatigue in Emergency Center Patients
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fatigue in Emergency Center Patients
Number analyzed (Participants) | 14
Age Continuous [Median (Full Range); unit: years] | 66 [28 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Patient Fatigue Severity Scores Assessed With MDASI
Description: Descriptive factor and cluster analysis using MD Anderson Symptom Index (MDASI) 13 core symptom items to form 1) treatment-related factor (nausea and vomiting) and 2) general severity factor (the remaining 11 core symptom items). Patients rate intensity and interference of symptoms on 0-10 numeric scales from "not present" to "as bad as you can imagine." Patients also rate the amount of interference with daily activities caused by symptoms on 0-10 numeric scales from "did not interfere" to "interfered completely."
Time Frame: Survey and blood draw done within 24 hours of patient's Emergency Center visit
Population: Study terminated early due to low recruitment, insufficient data for analysis.
Arm/Group | Fatigue in Emergency Center Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 Years
Arm/Group | Fatigue in Emergency Center Patients
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

LIMITATIONS AND CAVEATS:
Early termination led to small numbers of subjects, too little data to analyze.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No